CLINICAL TRIAL: NCT00594958
Title: Comparison of Three Batches of the Japanese Encephalitis Vaccine IC51. Double Blind, Randomized, Controlled Phase 3 Study.
Brief Title: Comparison of Three Batches of the Japanese Encephalitis Vaccine IC51
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IC51-309
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Results first posted 2014-01-23 (Estimated); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- IC51 Group A (Active Comparator): IC51 (JE-PIV) 6 mcg i.m. with 2 injections (days 0 and 28) with a vaccine produced from one out of three IC51 batches
  Interventions: Biological: IC51
- IC51 Group B (Active Comparator): IC51 (JE-PIV) 6 mcg i.m. with 2 injections (days 0 and 28) with a vaccine produced from one out of three IC51 batches
  Interventions: Biological: IC51
- IC51 Group C (Active Comparator): IC51 (JE-PIV) 6 mcg i.m. with 2 injections (days 0 and 28) with a vaccine produced from one out of three IC51 batches
  Interventions: Biological: IC51

INTERVENTIONS:
Biological: IC51 — 6 mcg, intramuscularly [i.m.], 0.5 mL
  Other Names: Japanese Encephalitis purified inactivated vaccine

SUMMARY:
The objective is to demonstrate equivalence of three IC51 batches in terms of Geometric Mean Titers for anti-JEV neutralizing antibody.

DETAILED DESCRIPTION:
This is a randomized, controlled, multi-center, double blind phase 3 study. The study population consists of male and female healthy subjects, aged at least 18 years.

624 subjects will be enrolled at approximately 6 sites in study centers in Austria and Germany.

ELIGIBILITY:
Main Inclusion Criteria:

* Male and female subjects aged at least 18 years with written informed consent and either no childbearing potential or negative pregnancy test

Main Exclusion Criteria:

* History of immunodeficiency or immunosuppressive therapy, known HIV, drug addiction including alcohol dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 639 (Actual)
Dates: Start 2006-09; Primary Completion 2007-04 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Eder, Mag., Study Director — Valneva Austria GmbH

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IC51 Group A | IC51 Group B | IC51 Group C
Started | 214 | 213 | 212
Randomized and at Least 1 Vaccination | 212 | 213 | 211
Completed | 200 | 210 | 202
Not Completed | 14 | 3 | 10
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Adverse Event | 4 | 1 | 2
Not completed — Pregnancy | 0 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 2
Not completed — Lost to Follow-up | 5 | 0 | 3
Not completed — administrative | 3 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety population, i.e. subjects who received at least one vaccination
Groups:
- Total: Total of all reporting groups
Arm/Group | IC51 Group A | IC51 Group B | IC51 Group C | Total
Number analyzed (Participants) | 212 | 213 | 211 | 636
Age, Continuous [Mean (Standard Deviation); unit: years] — numbers based on Safety Population: subjects with at least one vaccination
  years | 31.7 (10.8) | 31.3 (11.0) | 30.7 (10.3) | 31.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants] — numbers based on Safety Population: subjects with at least one vaccination
  Participants
    Female | 108 | 123 | 119 | 350
    Male | 104 | 90 | 92 | 286
Region of Enrollment [Number; unit: participants]
  Europe | 212 | 213 | 211 | 636

OUTCOME MEASURES:

1. Primary Outcome: GMT for Anti-JEV Neutralizing Antibody
Description: Equivalence between batches with regards to GMT (Geometric Mean Titer) was postulated if all three pair-wise 95 % Confidence Intervals for GMT ratios were between 0.5 and 2.
Time Frame: day 56
Population: Per Protocol Population (observed values)
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | IC51 Group A | IC51 Group B | IC51 Group C
Number analyzed (Participants) | 197 | 202 | 200
GMT | 160.71 [140.54 to 183.76] | 272.24 [237.22 to 312.43] | 127.56 [109.51 to 148.57]

2. Secondary Outcome: Safety
Description: Safety laboratory parameters, rate of SAEs and medically attended AEs, systemic and local tolerability
Time Frame: study duration
Reporting Status: Not Posted

3. Secondary Outcome: SCR for Anti-JEC Neutralizing Antibody Titer
Time Frame: day 56
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to Month 6
Arm/Group | IC51 Group A | IC51 Group B | IC51 Group C
Serious Adverse Events (participants affected / at risk) | 3/212 | 2/213 | 5/211
Other Adverse Events (participants affected / at risk) | 102/212 | 124/213 | 114/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IC51 Group A (N=212) | IC51 Group B (N=213) | IC51 Group C (N=211)
Reflux Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Acute Abdomen (Gastrointestinal disorders) | 0 | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 1
Peritonsillar Abscess (Infections and infestations) | 0 | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Intracranial Aneurysm (Nervous system disorders) | 1 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IC51 Group A (N=212) | IC51 Group B (N=213) | IC51 Group C (N=211)
Nausea (Gastrointestinal disorders) | 10 | 21 | 15
Fatigue (General disorders) | 21 | 30 | 34
Influenza Like Ilness (General disorders) | 24 | 35 | 32
Nasopharyngitis (Infections and infestations) | 28 | 34 | 30
Rhinitis (Infections and infestations) | 12 | 12 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 21 | 18
Headache (Nervous system disorders) | 42 | 51 | 52
Diarrhoea (Gastrointestinal disorders) | 2 | 5 | 4
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 3
Rash (Skin and subcutaneous tissue disorders) | 4 | 5 | 1
Acute Tonsillitis (Infections and infestations) | 5 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 7 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other